CLINICAL TRIAL: NCT04865614
Title: Comparison Between Inhalation and Intravenous Induction of Anaesthesia During Interventional Mitral Valve Repair
Acronym: COMPETENT
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Dr. Adrian Stephan, Principal Investigator, Heidelberg University
Other Study IDs: COMPETENT
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Blood Pressure; Hypotension Drug-Induced
MeSH Terms: conditions — Hypotension | interventions — Etomidate; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Etomidate group: Patients who received etomidate for induction of anaesthesia during interventional mitral valve repair (Mitraclip)
  Interventions: Drug: Etomidate
- Sevoflurane group: Patients who received sevoflurane for induction of anaesthesia during interventional mitral valve repair (Mitraclip)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Etomidate — Use of etomidate
  Groups: Etomidate group
Drug: Sevoflurane — Use of sevoflurane
  Groups: Sevoflurane group

SUMMARY:
The induction of anaesthesia is one of the most critical situations for high-risk-patients undergoing interventions surgery. For several reasons, it is crucial to maintain adequate blood pressure and cardiac output during this phase.

This retrospective cohort study aims to find out if the choice of the induction agent has a major impact on blood pressure and the use of catecholamines during the induction and the interventional procedure in patients undergoing interventional mitral valve repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective interventional mitral valve repair
* Sevoflurane or etomidate have been used for induction of anesthesia

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing interventional mitral valve repair
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Post-induction hypotension | First 20 minutes after induction of anaesthesia
  Hypotension in the first 20 minutes after induction of anesthesia

SECONDARY OUTCOMES:
Use of catecholamines after induction during the first 20 minutes after inductionafter induction | First 20 minutes after induction
  Use of catecholamines during the first 20 minutes after induction of anaesthesia
Use of catecholamines | Length of procedure (Approximately 60 to 90 minutes in average)
  Use of catecholamines during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adrian E Stephan, MD, Principal Investigator — Heidelberg University
Locations (1):
- Anästhesiologische Klinik (Universitätsklinikum Heidelberg), Heidelberg, Baden-Würtemberg, Germany

IPD SHARING:
Plan to Share IPD: No